CLINICAL TRIAL: NCT06665581
Title: Keratinocyte Skin Cancer Surgery in the Elderly, Aged 80 Years and Over, is Effective and Safe: a Single Institution Retrospective Study Over One Year
Brief Title: Keratinocyte Skin Cancer Surgery in the Elderly, Aged 80 Years and Over, is Effective and Safe
Status: Completed | Type: Observational
Sponsor: Juerg Hafner (Other)
Responsible Party: Sponsor-Investigator, Juerg Hafner, University Hospital Zurich, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: GerSurg
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
As a result of a longer life expectancy and a change in UV exposure, physicians will be facing a growing number of elderly patients with keratinocyte cancer (KC) in fair-skinned populations. The purpose of this study is to better characterize KC surgery in patients over 80 years and older with different comorbid conditions and to investigate the incidence of complications associated with KC surgery.

A retrospective monocentric study of patients aged 80 and older, having surgery for KC in University Hospital of Zurich between January 1, 2022, and December 31, 2022, was conducted. Demographics, comorbidities, current medication, treatment type, tumor characteristics, surgical defect size, repair type and complications within 6 months after surgery were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 80 and older, having surgery for KC in University Hospital of Zurich between January 1, 2022, and December 31, 2022

Exclusion Criteria:

* Presence of a documented rejection.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 80 and older having surgery for KC in University Hospital of Zurich between January 1, 2022, and December 31, 2022. All patients included in the study were operated on by the same dermatologic surgery team of University Hospital of Zurich under local anesthe-sia
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of complications associated with KC surgery in individuals aged 80 years and older | From January 1, 2022, to December 31, 2022

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Dermatology Clinic, Zurich, Canton of Zurich
  - University Hospital Zurich, Zurich, Canton of Zurich